CLINICAL TRIAL: NCT07054281
Title: UNITY VCS Vitreoretinal Surgery: Randomized Comparative Clinical Trial
Brief Title: UNITY VCS Vitreoretinal Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's business decision based on strategic shifts
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTV678-P001
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Epiretinal Membrane; Macular Hole; Visually Significant Vitreous Floater; Vitreomacular Traction; Vitreous Hemorrhage; Proliferative Diabetic Retinopathy; Rhegmatogenous Retinal Detachment; Retained Lens Material in the Posterior Segment
Keywords: Vitreoretinal Disease
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations; Vitreous Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- UNITY Vitreoretinal Cataract System (VCS) (Experimental): Vitreoretinal ophthalmic surgery in one eye using UNITY Vitreoretinal Cataract System (VCS)
  Interventions: Device: UNITY Vitreoretinal Cataract System (VCS); Procedure: Vitreoretinal ophthalmic surgery
- CONSTELLATION Vision System (Active Comparator): Vitreoretinal ophthalmic surgery in one eye using CONSTELLATION Vision System
  Interventions: Device: CONSTELLATION Vision System; Procedure: Vitreoretinal ophthalmic surgery

INTERVENTIONS:
Device: UNITY Vitreoretinal Cataract System (VCS) — UNITY VCS is a commercially approved surgical system that facilitates the management of fluid and gases, as well as removal, grasping, cutting, illumination, and coagulation of ocular materials during eye surgery. In this study, the UNITY VCS posterior segment functionalities will be used to perform posterior segment (i.e., vitreoretinal) ophthalmic surgery.
  Arms: UNITY Vitreoretinal Cataract System (VCS)
Device: CONSTELLATION Vision System — CONSTELLATION is a commercially approved, multifunctional surgical instrument used during ophthalmic surgery to cut vitreous and tissues, emulsify the lens, illuminate the posterior segment of the eye, and apply diathermy to stop bleeding.
  Arms: CONSTELLATION Vision System
Procedure: Vitreoretinal ophthalmic surgery — Ophthalmic surgery performed in the posterior segment of the eye

SUMMARY:
This purpose of this study is to compare the safety and effectiveness of two eye surgery systems-UNITY VCS and CONSTELLATION-in treating adults with vitreoretinal diseases or disorders.

DETAILED DESCRIPTION:
Subjects will attend a total of 6 scheduled visits for an individual of participation of approximately 3 months. One eye (study eye) will be treated with either UNITY VCS or CONSTELLATION, as randomized.

ELIGIBILITY:
Key Inclusion Criteria:

* Requires surgery for a clinically documented posterior vitreoretinal medical condition.
* Clear ocular media except for vitreous hemorrhage and floaters undergoing surgery.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Presence of clinically significant ocular or systemic diseases that may interfere with study outcomes or safety.
* Diagnosis of glaucoma or suspected ocular hypertension.
* Recent intraocular eye surgery, other than cataract surgery, resulting in retained lens materials in the posterior segment (within the past 3-months).
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of vitreoretinal surgeries performed using 27-gauge consumables | Day 0 operative
  The surgeon will select the gauge size of the surgical consumables used for vitreoretinal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Retina Associates of Orange County, Laguna Hills, California
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - NYC Retina - Manhattan, New York, New York
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Charles Retina Institute, Germantown, Tennessee
  - The Eye Institute of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No